CLINICAL TRIAL: NCT05771922
Title: Role of New High Resolution Ultrasonographic Modalities for Diagnosis of Fetal Nervous System Anomalies
Brief Title: Implication of New High Resolution Ultrasonographic Modalities for Diagnosis of Fetal Nervous System Anomalies
Status: Recruiting | Type: Observational
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Professor Atef Darwish, Senior consultant of Obstetrics and Gynecology, Woman's Health University Hospital, Egypt
Other Study IDs: 1234567
Record Dates: First submitted 2023-03-05; First posted 2023-03-16 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Ultrasound Therapy; Complications Anomaly Central Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: High-resolution ultrasonography — High-resolution ultrasonography to detect fetal CNS anomalies

SUMMARY:
The fetal CNS screening examination during the mid-trimester scan in low-risk pregnancies should include evaluation of the fetal head and spine, using transabdominal sonography. Evaluation of two axial planes allows visualization of the relevant cerebral structures to assess the anatomic integrity of the fetal brain.These planes are commonly referred to as the transventricular and transcerebellar planes. A third plane, the so-called transthalamic plane, is frequently added, mostly for the purpose of biometry. Structures that should be noted in the routine examination include the lateral ventricles, the cerebellum, the cisterna magna, and the cavum septi pellucidi (CSP). Head shape and brain texture should also be noted on these views.

DETAILED DESCRIPTION:
The neural system malformation is one of the more common congenital anomalies encountered in pregnancy. They represent about 0.3-1 percent of all live births. During a prenatal anomaly scan, detection of CNS malformations is important, especially since these anomalies have a poor prognosis and are also associated with genetic syndromes or chromosomal anomalies. Such malformations have clinical importance because they are associated with high rates of morbidity and mortality, influencing the neurocognitive and motor development of the survivors, who may have lifelong sequelae. Thus, it's extremely important to assess the fetal CNS during the prenatal period in order to identify any changes in its development and give appropriate advice to parents regarding pregnancy follow-up. Also, it is vital to explore options for fetal therapy and the timing/type of delivery, as well as postnatal treatment and prognosis.

The fetal CNS screening examination during the mid-trimester scan in low-risk pregnancies should include evaluation of the fetal head and spine, using transabdominal sonography. Evaluation of two axial planes allows visualization of the relevant cerebral structures to assess the anatomic integrity of the fetal brain.These planes are commonly referred to as the transventricular and transcerebellar planes. A third plane, the so-called transthalamic plane, is frequently added, mostly for the purpose of biometry. Structures that should be noted in the routine examination include the lateral ventricles, the cerebellum, the cisterna magna, and the cavum septi pellucidi (CSP). Head shape and brain texture should also be noted on these views.

ELIGIBILITY:
Inclusion Criteria:

Suspicion of CNS or spinal malformation at routine screening ultrasound Suspicion of CNS or spinal malformation at nuchal translucency scan Family history of inheritable CNS spinal malformations Previous pregnancy complicated by fetal brain or spinal malformation Fetus with congenital heart disease Monochorionic twins Suspected congenital intrauterine infection Exposure to teratogens known to affect neurogenesis

Exclusion Criteria:

Low risk pregnancy

Ages: 20 Years to 28 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: all pregnant women with gestational age between 20 and 28 weeks coming to outpatient clinic for antenatal care with one or more of the following inclusion criteria will be included in this study.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
PREVELANCE OF FETAL BRAIN ANOMALIES UTILIZING THREE-AXIAL VIEW WITH 2D ULTRASONOGRAPHY | 2 years
  tO DETECT PREVELANCE OF FETAL BRAIN CONGENITAL ANOMALIES UTILIZING STANDARD THREE-AXIAL VIEW (TRANSTHALAMIC, TRANSVENTRICULAR AND TRANSCEREBELLER ) WITH 2D ULTRASONOGRAPHY
PREVELANCE OF FETAL BRAIN ANOMALIES UTILIZING ADDITIONAL 2 VIEWS TO THE STANDARD THREE-AXIAL VIEW WITH 2D ULTRASONOGRAPHY | 2 years
  PREVELANCE OF FETAL BRAIN ANOMALIES UTILIZING ADDITIONAL 2 VIEWS (TRANCALVERIAL AND TRANSGENU AND SPELNIUM) TO THE STANDARD THREE-AXIAL VIEW WITH 2D ULTRASONOGRAPHY .
PREVELANCE OF FETAL NERVOUS SYSTEM ANOMALIES UTILIZING 3D ULTRASONOGRAPHY . | 2 years
  PREVELANCE OF FETAL NERVOUS SYSTEM ANOMALIES UTILIZING 3D ULTRASONOGRAPHY BY SURFACE 3 D, MULTIPLANNER AND MULTISLICE VIEWS .

CONTACTS AND LOCATIONS:
Locations (1):
- Woman's Health University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided